CLINICAL TRIAL: NCT04084561
Title: Nicotine Dependence and Lung Cancer Genetics in African Americans
Brief Title: Risk Communication in African American Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-8004; 1U54CA221705-01A1 (NIH)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRHA (Experimental): High Risk, High Ancestry
  Interventions: Behavioral: HRHA
- LRLA (Experimental): Low Risk, Low Ancestry
  Interventions: Behavioral: LRLA
- HRLA (Experimental): High Risk, Low Ancestry
  Interventions: Behavioral: HRLA
- LRHA (Experimental): Low Risk, High Ancestry
  Interventions: Behavioral: LRHA

INTERVENTIONS:
Behavioral: HRHA — participants will be asked to consider a hypothetical scenario in which genetic test results reveal that: 1) they carry genotypes that place African American smokers at a particularly high (~50%-80%) risk for the development of lung cancer, and 2) their genetic profile reflects a particularly high concordance with African heritage (~90%).
  Arms: HRHA
Behavioral: LRLA — participants will be asked to consider a scenario in which genetic test results reveal that: 1) they are at normal (~7%-10%) risk for the development of lung cancer, and 2) their genetic profile reflects a particularly low concordance with African heritage (~10%).
  Arms: LRLA
Behavioral: HRLA — participants will receive "High Risk, Low Ancestry (HRLA)" hypothetical
  Arms: HRLA
Behavioral: LRHA — participants will receive "Low Risk, High Ancestry (HRLA)" hypothetical
  Arms: LRHA

SUMMARY:
The study aims to understand the effects of learning about one's genetic risk for lung cancer that is specific to their ancestry. Participants will be given hypothetical personalized genetic risk results and ask to think about how they might respond to such information if they actually received such results.

DETAILED DESCRIPTION:
The study aims to understand the effects of learning about one's genetic risk for lung cancer that is specific to their ancestry. Smokers will be randomized to receive hypothetical information about their genetic status and consider how they think they would respond if such results were actually presented to them. They will be randomly assigned to receive one of four sets of hypothetical genetic results: 1) High risk of lung cancer and high genetic African ancestry, 2) High risk of lung cancer and low genetic African ancestry, 3) Low risk of lung cancer and high genetic African ancestry, or 4) Low risk of lung cancer and low genetic African ancestry. After being given this hypothetical information, participants will complete brief questionnaires assessing perceived risk of lung cancer, worry about cancer, psychological distress, and motivation to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age minimum
* Self-report African American
* Report smoking at least 100 lifetime cigarettes

Exclusion Criteria:

* Report history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Ragin, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Hunter College, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because of COVID, and with the consent of the funding agency and IRB, we opened a second IRB to JUST do Aim 3. So Aim 3 is independent and it is the only part that was a clinical trial. This sample consisted of 166 respondents.
Pre-assignment Details: Aim3 was the clinical trial component. We were initially informed by clinical trials staff that we should include enrollment numbers for ALL of the aims. Then we were informed to include only those recruited to Aim 3. Although the original goal was to recruit participants from Aims 1 and 2 to do Aim 3, COVID-19 made that impossible. Thus, with consent of the funding agency and IRB, we pivoted to collect the Aim 3 data remotely in an independent sample. This sample consisted of 166 respondents.
Period: Overall Study
Arm/Group | HRHA | LRLA | HRLA | LRHA
Started | 41 | 40 | 43 | 42
Completed | 41 | 40 | 43 | 42
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRHA | LRLA | HRLA | LRHA | Total
Number analyzed (Participants) | 41 | 40 | 43 | 42 | 166
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.80 (13.478) | 43.24 (13.821) | 41.58 (15.462) | 37.62 (14.629) | 41.28 (14.428)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 25 | 27 | 102
  Male | 15 | 16 | 18 | 15 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Americans | 41 | 40 | 43 | 42 | 166

OUTCOME MEASURES:

1. Primary Outcome: Motivation to Quit Smoking
Description: use self report 7 item (condition options) MTSS (Motivation to Stop Smoking) Scale with yes/no option to determine the quitting intention condition; range of scale : 1-7, with higher score means higher motivation to quit smoking
Time Frame: 1 minute after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HRHA | LRLA | HRLA | LRHA
Number analyzed (Participants) | 41 | 40 | 43 | 42
units on a scale | 4.95 (.296) | 3.30 (.254) | 5.49 (.261) | 4.52 (.284)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | HRHA | LRLA | HRLA | LRHA
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/43 | 0/42

LIMITATIONS AND CAVEATS:
This study examined the effects of communicating hypothetical genetic results to patients on their motivation to quit smoking. Future research needs to study effects of actual genetic risk communication, and its effects on actual smoking cessation behavior, rather than motivation to quit. Nevertheless the results suggest communicating elevated risk of lung cancer may increase motivation to quit smoking.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT04084561/Prot_SAP_000.pdf